CLINICAL TRIAL: NCT06279910
Title: Inclusion of Calcifediol in the Hospital Therapeutic Protocol for Treatment of SARS-CoV-2 Disease (COVID-19). Mortality Analysis. Retrospective Study.
Brief Title: Calcifediol in the Treatment of SARS-CoV-2 Disease (COVID-19).
Acronym: COVIDIOL
Status: Completed | Type: Observational
Sponsor: Complejo Hospitalario Universitario de Albacete (Other)
Responsible Party: Sponsor
Other Study IDs: 2021 36 (EOm)
Record Dates: First submitted 2024-02-25; First posted 2024-02-28 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: SARS-CoV 2 Pneumonia
Keywords: Calcifediol; Cathelicidin peptide; Corticoids; COVID-19; Cytokine storm; Multiorgan failure; Pneumonia; Respiratory distress syndrome (ARDS); Respiratory failure; SARS-CoV-2; Vitamin D; Vitamin D endocrine system; VDR Vitamin D
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Multiple Organ Failure; Pneumonia; Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — Calcifediol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Patients treated with calcifediol: Patients admitted to the CHUA, due to COVID-19 [respiratory infection confirmed by radiographic pattern of viral pneumonia and positive polymerase chain reaction (PCR)/antigen for SARS-CoV-2] treated with calcifediol
  Interventions: Drug: Calcifediol
- Patients not treated with calcifediol: Patients admitted to the CHUA, due to COVID-19 (respiratory infection confirmed by radiographic pattern of viral pneumonia and positive PCR/antigen for SARS-CoV-2) not treated with calcifediol

INTERVENTIONS:
Drug: Calcifediol — Calcifediol added as a treatment to the rest of the prescribed drugs of the protocol
  Groups: Patients treated with calcifediol

SUMMARY:
Descriptive, retrospective, observational, anonymous, study to evaluate the potential effect of incorporating calcifediol into the therapeutic protocol of patients hospitalized for COVID-19 on mortality and other outcome variables, such as admission to the Intensive Care Unit (ICU), to "Complejo Hospitalario Universitario de Albacete" (CHUA). Albacete (Spain)", based on the files of the MXXI medical records, Information System of the Laboratory (ISL) and Pharmacy.

DETAILED DESCRIPTION:
The coronavirus disease-19 (COVID-19) pandemic, caused by the severe acute respiratory syndrome β-coronavirus (SARS-CoV-2), is one of the greatest challenges facing modern medicine and public health systems worldwide. Since its appearance in December 2019, it has caused nearly 7 million deaths, recognized, and confirmed worldwide, with high acute and post-acute morbidity, making it one of the deadliest in human history, with a devastating impact on national economies worldwide.

In the first outbreaks of COVID-19, although 80% were asymptomatic or had mild symptoms, 20% of patients developed severe symptoms, and 5% presented acute respiratory distress syndrome (ARDS), septic shock and accompanied multi-organ organ failure, with a high risk of death. Numerous risk factors have been described that influence the poor outcome of these patients, such as age, sex, high blood pressure, chronic obstructive pulmonary disease, diabetes, obesity, chronic lung and digestive diseases, asthma, chronic heart disease, cancer, D-dimer greater than 1000, or a high SOFA (Sequential Organ Failure Assessment Score). It has also been observed that patients with no a priori risk factors may have a poor outcome.

The scientific community immediately proposed strong social containment measures, quickly developed effective vaccines to prevent the appearance of severe clinical forms of COVID-19, and developed new treatments against all aspects of the disease: antiviral agents, anti-inflammatory agents, antithrombotic therapies, therapies against hypoxemic acute respiratory failure, therapies with anti-SARS-CoV-2 antibodies (neutralizing), modulators of the renin-angiotensin-aldosterone system and vitamins, so that social and economic activity has gradually recovered worldwide.

However, at the current time, there are some indications that hospital admissions for COVID-19 are on the rise again, so the pandemic seems far from over and future waves of infection are likely. These indications update and highlight again the repositioning strategy used since the beginning of the pandemic for the use of safe drugs, approved for another indication, and redirected to improve symptoms and clinical outcomes in patients with COVID-19. Various drugs have been investigated under this strategy and many studies have been published, some of them successful.

In this sense, during the first months of the pandemic, on the basis of biological plausibility, the investigators thought that the activation of the vitamin D receptor (VDR) signaling pathway of the vitamin D endocrine system (VDES) could produce beneficial effects in COVID-19. These effects were achieved by improving innate antiviral effector mechanisms, facilitating the induction of antimicrobial peptides/autophagy, mitigating the subsequent reactive hyperinflammatory phase of the host, decreasing the cytokine/chemokine storm, modulating the expression of the renin angiotensin system (RAAS) and neutrophil activity, maintaining the integrity of the pulmonary/intestinal epithelial barrier, stimulating epithelial repair and directly and indirectly reducing the increase in coagulability and prothrombotic tendency associated with a severe course of COVID-19 and its complications. Available evidence suggests that VDES/VDR stimulation, while maintaining optimal serum 25-hydroxyvitamin D [(25(OH)D)] status, in patients with SARS-CoV-2 infection may significantly reduce the risk of distress syndrome, acute respiratory distress syndrome (ARDS) and the development of severe COVID-19.

The investigators decided to use calcifediol, which is a prohormone (and cornerstone of the VDES) and substrate for the synthesis of the system's hormone, calcitriol. The poor availability of calcifediol described in the general population, most marked in patients affected by COVID, means that the potential protection that VDR/VDES stimulation confers against various aspects of the disease is lost.

Calcifediol provides pharmacokinetic advantages, which give it a certain functional superiority over native vitamin D3 and even over the hormonal form of VDES, calcitriol, for its use in COVID-19. It is very hydrophilic and, therefore, after oral ingestion, it is absorbed through the portal venous system and does not require hydroxylation at the 25 position, immediately increasing optimal circulating concentrations of 25(OH)D3. Therefore, even if administered orally, it is available at high concentrations within a few hours, and in a stable manner, to be a substrate for calcitriol synthesis at the kidney and other target organs in COVID-19.

The clinical trial pilot study and several observational intervention studies using relatively high doses of calcifediol (0.532 µg on day 1 and 0.266 µg on days 3, 7, 14, 21 and 28) decreased the severity of the disease, dramatically reducing the need for ICU admission, severity, and mortality rate.

Therefore, using calcifediol at the doses described for rapid correction of 25(OH)D deficiency in all patients in the early stages of COVID-19, in association with the best available therapy, was assessed as a good option for the treatment of COVID-19. For this reason, on January 24, 2021, the CHUA incorporated calcifediol into the protocol "Recommendations for action and treatment of the coronavirus SARS-CoV-2 disease" (COVID-19) version 11.1".

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the hospital CHUA
2. Meet the SARS-CoV-2 diagnostic criteria with positive PCR
3. They have completed at least the first dose of Calcifediol within the first 72 hours after admission, (according to protocol).

Exclusion Criteria:

1. Patients who do not receive the full first dose of Calcifediol within the first 72 hours.
2. Patients for whom electronic medical record data cannot be collected.
3. Patients with other serious intercurrent diseases (eg advanced oncological pathology).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the CHUA, due to COVID-19 [respiratory infection confirmed by radiographic pattern of viral pneumonia and positive PCR/antigen for SARS-CoV-2]. Those participants for whom there is not enough information in the files to be able to analyze the study hypotheses will be excluded from the study.
  Patients meeting ALL inclusion criteria and NO exclusion criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Measure mortality by differentiating groups: calcifediol yes/no. | 02/21/2024 to 04/25/2024
  Measure mortality by differentiating groups: calcifediol yes/no.
Measure the need for ICU admission by differentiating the groups calcifediol yes/no. | 02/21/2024 to 04/25/2024
  Measure the need for ICU admission by differentiating the groups calcifediol yes/no.

SECONDARY OUTCOMES:
Measure mortality in relation to baseline 25(OH)D levels | 02/21/2024 to 04/25/2024
  Measure mortality in relation to baseline 25(OH)D levels
To evaluate the effect of calcifediol treatment on mortality in patients with severe 25(OH)D deficiency | 02/21/2024 to 04/25/2024
  To evaluate the effect of calcifediol treatment on mortality in patients with severe 25(OH)D deficiency
Measure the composite variable poor prognosis, (death and ICU) by differentiating the groups calcifediol yes/no | 02/21/2024 to 04/25/2024
  Measure the composite variable poor prognosis, (death and ICU) by differentiating the groups calcifediol yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Javier Torres, PhD, Study Chair — Complejo Hospitalario Universitario de Albacete. Albacete. Spain; Jose M Quesada, MD, Study Director — Maimónides Biomedical Research Institute of Córdoba (IMIBIC). Córdoba. Spain
Locations (1):
- Complejo Hospitalario Universitario de Albacete, Albacete, Albacete, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymized information collected from patients will be shared publicly upon request. All information related to variables or results included in the study will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available in the following months after all results will have been published.
Access Criteria: All data requests will be reviewed by the principal investigator of the project. Data will be shared upon reasonable request to be examined or reviewed. It will not be permitted to carry out any other kind of study (including statistical) by people other than the researchers of the main study.

REFERENCES:
- [Background] Ranabhat CL, Jakovljevic M, Kim CB, Simkhada P. COVID-19 Pandemic: An Opportunity for Universal Health Coverage. Front Public Health. 2021 Jul 29;9:673542. doi: 10.3389/fpubh.2021.673542. eCollection 2021. No abstract available. PMID 34395361
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Bowe B, Xie Y, Al-Aly Z. Postacute sequelae of COVID-19 at 2 years. Nat Med. 2023 Sep;29(9):2347-2357. doi: 10.1038/s41591-023-02521-2. Epub 2023 Aug 21. PMID 37605079
- [Background] Giliberto Capano, Michael Howlett, Darryl S L Jarvis, M Ramesh, Long-term policy impacts of the coronavirus: normalization, adaptation, and acceleration in the post-COVID state, Policy and Society, 2022; 41 (1): 1-12, doi: 10.1093/polsoc/puab018
- [Background] Wiersinga WJ, Rhodes A, Cheng AC, Peacock SJ, Prescott HC. Pathophysiology, Transmission, Diagnosis, and Treatment of Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 Aug 25;324(8):782-793. doi: 10.1001/jama.2020.12839. PMID 32648899
- [Background] Pritchard E, Matthews PC, Stoesser N, Eyre DW, Gethings O, Vihta KD, Jones J, House T, VanSteenHouse H, Bell I, Bell JI, Newton JN, Farrar J, Diamond I, Rourke E, Studley R, Crook D, Peto TEA, Walker AS, Pouwels KB. Impact of vaccination on new SARS-CoV-2 infections in the United Kingdom. Nat Med. 2021 Aug;27(8):1370-1378. doi: 10.1038/s41591-021-01410-w. Epub 2021 Jun 9. PMID 34108716
- [Background] Murakami N, Hayden R, Hills T, Al-Samkari H, Casey J, Del Sorbo L, Lawler PR, Sise ME, Leaf DE. Therapeutic advances in COVID-19. Nat Rev Nephrol. 2023 Jan;19(1):38-52. doi: 10.1038/s41581-022-00642-4. Epub 2022 Oct 17. PMID 36253508
- [Background] El-Sadr WM, Vasan A, El-Mohandes A. Facing the New Covid-19 Reality. N Engl J Med. 2023 Feb 2;388(5):385-387. doi: 10.1056/NEJMp2213920. Epub 2023 Jan 28. No abstract available. PMID 36724378
- [Background] The Lancet. The COVID-19 pandemic in 2023: far from over. Lancet. 2023 Jan 14;401(10371):79. doi: 10.1016/S0140-6736(23)00050-8. No abstract available. PMID 36641201
- [Background] Kato Y, Nishiyama K, Nishimura A, Noda T, Okabe K, Kusakabe T, Kanda Y, Nishida M. Drug repurposing for the treatment of COVID-19. J Pharmacol Sci. 2022 Jul;149(3):108-114. doi: 10.1016/j.jphs.2022.04.007. Epub 2022 Apr 25. PMID 35641023
- [Background] Quesada-Gomez JM, Entrenas-Castillo M, Bouillon R. Vitamin D receptor stimulation to reduce acute respiratory distress syndrome (ARDS) in patients with coronavirus SARS-CoV-2 infections: Revised Ms SBMB 2020_166. J Steroid Biochem Mol Biol. 2020 Sep;202:105719. doi: 10.1016/j.jsbmb.2020.105719. Epub 2020 Jun 11. PMID 32535032
- [Background] Quesada-Gomez JM, Lopez-Miranda J, Entrenas-Castillo M, Casado-Diaz A, Nogues Y Solans X, Mansur JL, Bouillon R. Vitamin D Endocrine System and COVID-19: Treatment with Calcifediol. Nutrients. 2022 Jun 29;14(13):2716. doi: 10.3390/nu14132716. PMID 35807895
- [Background] Quesada-Gomez JM, Bouillon R. Calcifediol Cornerstone of the Vitamin D Endocrine System. Nutrients. 2023 May 12;15(10):2290. doi: 10.3390/nu15102290. PMID 37242173
- [Background] Lips P, Cashman KD, Lamberg-Allardt C, Bischoff-Ferrari HA, Obermayer-Pietsch B, Bianchi ML, Stepan J, El-Hajj Fuleihan G, Bouillon R. Current vitamin D status in European and Middle East countries and strategies to prevent vitamin D deficiency: a position statement of the European Calcified Tissue Society. Eur J Endocrinol. 2019 Apr;180(4):P23-P54. doi: 10.1530/EJE-18-0736. PMID 30721133
- [Background] Wang Z, Joshi A, Leopold K, Jackson S, Christensen S, Nayfeh T, Mohammed K, Creo A, Tebben P, Kumar S. Association of vitamin D deficiency with COVID-19 infection severity: Systematic review and meta-analysis. Clin Endocrinol (Oxf). 2022 Mar;96(3):281-287. doi: 10.1111/cen.14540. Epub 2021 Jul 12. PMID 34160843
- [Background] Bouillon R, Quesada-Gomez JM. Vitamin D Endocrine System and COVID-19. JBMR Plus. 2021 Nov 17;5(12):e10576. doi: 10.1002/jbm4.10576. eCollection 2021 Dec. PMID 34950831
- [Background] Bouillon R, Quesada Gomez JM. Comparison of calcifediol with vitamin D for prevention or cure of vitamin D deficiency. J Steroid Biochem Mol Biol. 2023 Apr;228:106248. doi: 10.1016/j.jsbmb.2023.106248. Epub 2023 Jan 13. PMID 36646151
- [Background] Entrenas Castillo M, Entrenas Costa LM, Vaquero Barrios JM, Alcala Diaz JF, Lopez Miranda J, Bouillon R, Quesada Gomez JM. "Effect of calcifediol treatment and best available therapy versus best available therapy on intensive care unit admission and mortality among patients hospitalized for COVID-19: A pilot randomized clinical study". J Steroid Biochem Mol Biol. 2020 Oct;203:105751. doi: 10.1016/j.jsbmb.2020.105751. Epub 2020 Aug 29. PMID 32871238
- [Background] Nogues X, Ovejero D, Pineda-Moncusi M, Bouillon R, Arenas D, Pascual J, Ribes A, Guerri-Fernandez R, Villar-Garcia J, Rial A, Gimenez-Argente C, Cos ML, Rodriguez-Morera J, Campodarve I, Quesada-Gomez JM, Garcia-Giralt N. Calcifediol Treatment and COVID-19-Related Outcomes. J Clin Endocrinol Metab. 2021 Sep 27;106(10):e4017-e4027. doi: 10.1210/clinem/dgab405. PMID 34097036
- [Background] Alcala-Diaz JF, Limia-Perez L, Gomez-Huelgas R, Martin-Escalante MD, Cortes-Rodriguez B, Zambrana-Garcia JL, Entrenas-Castillo M, Perez-Caballero AI, Lopez-Carmona MD, Garcia-Alegria J, Lozano Rodriguez-Mancheno A, Arenas-de Larriva MDS, Perez-Belmonte LM, Jungreis I, Bouillon R, Quesada-Gomez JM, Lopez-Miranda J. Calcifediol Treatment and Hospital Mortality Due to COVID-19: A Cohort Study. Nutrients. 2021 May 21;13(6):1760. doi: 10.3390/nu13061760. PMID 34064175